CLINICAL TRIAL: NCT03130556
Title: A Phase 1, Randomized, Open-label Study Of Glasdegib (Pf-04449913) In Healthy Volunteers To Establish The Bioequivalence Of The Phase 2 Formulation To The Glasdegib Ich Formulation And To Estimate The Potential Effect Of Food And A Proton Pump Inhibitor On Glasdegib Plasma Pharmacokinetics
Brief Title: A Study Of Glasdegib In Healthy Volunteers To Establish The Bioequivalence Of The Phase 2 Formulation To The ICH Formulation
Acronym: B1371026
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B1371026
Record Dates: First submitted 2017-04-21; First posted 2017-04-26 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Healthy Volunteers
Keywords: Glasdegib; PF-04449913; Pharmacokinetics; Bioavailability
MeSH Terms: interventions — glasdegib; Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Glasdegib BE and Food (Experimental): Subjects receive 100 mg single dose of ICH glasdegib under fasted condition with washout and then 100 mg single dose of Phase 2 tablet under fasted condition with washout in a randomized fashion. Finally subjects receive a 100 mg single dose ICH tablet after a high fat, high calorie meal.
  Interventions: Drug: Glasdegib; Other: High Fat, High Calorie Meal
- Glasdegib BE and PPI Effect (Experimental): Subjects receive 100 mg single dose of ICH glasdegib under fasted condition with washout and then 100 mg single dose of Phase 2 tablet under fasted condition with washout in a randomized fashion. Finally subjects receive a 100 mg single dose ICH tablet in the fasted state after repeated daily dosing with rabeprazole.
  Interventions: Drug: Glasdegib; Drug: Rabeprazole

INTERVENTIONS:
Drug: Glasdegib — Subjects receive 100 mg single dose of ICH glasdegib under fasted condition with washout and then 100 mg single dose of Phase 2 tablet under fasted condition with washout in a randomized fashion. Finally subjects either receive a 100 mg single dose ICH tablet after a high fat, high calorie meal or receive a 100 mg single dose of ICH tablet after repeated daily dosing with rabeprazole.
Other: High Fat, High Calorie Meal — A subset of subjects in the study will receive a high fat, high calorie meal prior to being administered a single 100 mg tablet ICH tablet of glasdegib.
  Arms: Glasdegib BE and Food
Drug: Rabeprazole — A subset of subjects will receive repeated daily dosing of 40 mg rabeprazole for 7 days with 100 mg single dose of ICH glasdegib being administered on Day 7.
  Arms: Glasdegib BE and PPI Effect

SUMMARY:
This study is intended to establish the bioequivalence (BE) of single 100 mg doses of glasdegib administered under fasted conditions to healthy volunteers as the ICH formulation compared to the Phase 2 formulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non-child bearing potential who, at the time of screening, are between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG or clinical laboratory tests. Female subjects of nonchildbearing potential must meet at least 1 of the following criteria:

  1. Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 24 consecutive months with no alternative pathological or physiological cause; with a serum follicle-stimulating hormone (FSH) level confirming the postmenopausal state;
  2. Have undergone a documented hysterectomy and/or bilateral oophorectomy;
  3. Have medically confirmed ovarian failure. All other female subjects (including females with tubal ligations and females that do NOT have a documented hysterectomy, bilateral oophorectomy and/or ovarian failure) are considered to be of childbearing potential.
* Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study. -. Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* A positive urine drug test.
* Screening supine 12-lead ECG demonstrating a corrected QT (QTc) interval >450 msec or a QRS interval >120 msec. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTc or QRS values should be used to determine the subject's eligibility.
* Subjects with family history of myocardial infarction, congenital long QT syndrome, torsades de pointes or clinically significant ventricular arrhythmias. Subjects should be within normal range of potassium, magnesium and corrected calcium calculation at screening.
* Pregnant female subjects; breastfeeding female subjects; female subjects of childbearing potential; male subjects with partners currently pregnant; male subjects who are unwilling or unable to use two highly effective methods of contraception as outlined in this protocol for the duration of the study and for at least 90 days after the last dose of investigational product and, refrain from sperm donation for the duration of the Study and for at least 90 days after the last dose of investigational product.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-07-06 (Actual); Study Completion 2017-07-21 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 5 days
Area Under the Curve From Time Zero to Last Measured Time Point [AUC (0 - t)] | 5 days

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Shaik N, Hee B, Wei H, LaBadie RR. Evaluation of the effects of formulation, food, or a proton-pump inhibitor on the pharmacokinetics of glasdegib (PF-04449913) in healthy volunteers: a randomized phase I study. Cancer Chemother Pharmacol. 2019 Mar;83(3):463-472. doi: 10.1007/s00280-018-3748-8. Epub 2018 Dec 10. PMID 30536154
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1371026&StudyName=A+Phase+1%2C+Randomized%2C+Open-label+Study+Of+Glasdegib+%28pf-04449913%29+In+Healthy+Volunteers+To+Establish+The+Bioequivalence+Of+The+Phase+2+Formulation+To+The+Glasdegib+Ich+Formulation+And+To+Estimate+The+Potential+Effect+Of+Food+And+A+Proton+Pump+Inhibitor+On+Glasdegib+Plasma+Pharmacokinetics